CLINICAL TRIAL: NCT03358992
Title: Clinical Evaluation for Sarcoma Originated From Bone
Acronym: CESOFB
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: Xijing Hospital (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: CBTRA-01
Record Dates: First submitted 2017-11-27; First posted 2017-12-02 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Sensitivity; Specificity; Histological Response; Survival
Keywords: CESOFB; clinical evaluation; RECIST; histological response; survival; osteosarcoma; Ewing sarcoma
MeSH Terms: conditions — Hypersensitivity; Osteosarcoma; Sarcoma, Ewing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Response Evaluation Criteria in Solid Tumors (RECIST) are insensitive in evaluating primary sarcoma originated from bone treated with chemotherapy or targeted therapy, which did not have the definition of measurement methods either. This study evaluates whether clinical imaging findings of sarcoma after preoperative chemotherapy correlate with tumor responses by pathological evaluation by Huvos classifications and develops reliable, quantitative, clinical response criteria.

DETAILED DESCRIPTION:
A total of 1570 lesions were evaluated by clinical imaging including X-ray, computed tomography, magnetic resonance imaging and bone scan or PET/CT preoperatively treated with chemotherapy. All patients had surgery in our center and get pathological evaluation by tumor necrosis rate. Statistical diversity analysis was performed by different pathological groups and Receiver Operating Characteristic Curves，ROC were done to find the dividing clinical parameters (Cut-off values) to distinguish different pathological groups.The cut-off values of change rate of maximum diameters of tumor located in extremities were 86%, 50.7% and 0.02% for Huvos Ⅳ,Ⅲ,ⅡandⅠgroups. The differentiation was not obvious using bone scan to distinguish different pathological responses. And the cut-off value for SUVmax value for Huvos Ⅲ,ⅡandⅠgroups were 60.7% and 31.4%.After Multidisciplinary discussion in multiple sites of China, we finally designed a evaluation system based on our data. This study is desgined to prospectively compare the sensitivity and specificity of this Clinical evaluation of primary sarcoma originated from bone with other clinical evaluation system,such as RECIST 1.1, Choi and PERCIST.

ELIGIBILITY:
Inclusion Criteria:

* 1) histologically confirmed high-grade osteosarcoma;
* 2) initially treated in Musculoskeletal Tumor Center of Peking University People's Hospital, Xijing Hospital or The Second Hospital affiliated to Zhejiang Hospital;
* 3) imaging evaluation should be available;
* 4) completed neo-adjuvant chemotherapy and at least 8 cycles of adjuvant chemotherapy;
* 5) expected to live longer than 3 months with Eastern Cooperative Oncology Group performance status of 0 or 1;
* 6) acceptable hematologic, hepatic, and renal function.

Exclusion Criteria:

* 1) Patients who could not complete neo-adjuvant chemotherapy or at least 4-month adjuvant chemotherapy;
* 2) lost to follow-up.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Biopsy proved high-grade osteosarcoma, who could follow routine chemo-protocol for osteosarcoma, could get enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12-30 (Estimated); Study Completion 2019-03-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | 12 months
  Sensitivity is defined as the true right clinical evaluated number/ the pathological evaluated number by different classification system.
Specificity | 12 months
  Specificity is defined as the true wrong clincial evuluated number /the pathological evaluated number by different classification system.
Pathological response rate | 12 months
  tumor necrosis rate descripted by Huvos

SECONDARY OUTCOMES:
progression-free survival | 24 months
  Progression-free survival is defined as time from diagnosis to the first occurrence of progression of disease or death from any cause
overall survival | 60 months
  overall survival is defined as time from diagnosis to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Guo, Principal Investigator — Musculoskeletal Tumor Center of Peking University People's Hospital
Locations (3):
- China (3):
  - The second affliated Hospital of Zhejiang University School of medicine, Hangzhou, Zhejiang
  - Musculoskeletal Tumor Center of Peking University People's Hospital, Beijing
  - Xijing Hospital, Xi'an

IPD SHARING:
Plan to Share IPD: Undecided